CLINICAL TRIAL: NCT05266430
Title: A Prospective Group-Matched Study of Visual Outcomes in Subjects Treated With Belzupacap Sarotalocan (AU-011) or Plaque Radiotherapy for Primary Indeterminate Lesions or Choroidal Melanoma (IL/ CM)
Brief Title: Prospective Group-Matched Study With Belzupacap Sarotalocan (Bel-sar; AU-011) or Plaque Radiotherapy for Primary Indeterminate Lesions or Choroidal Melanoma (IL/ CM)
Acronym: IL
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision - Low Enrollment
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: AU-011-402
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Choroidal Melanoma; Indeterminate Lesions
Keywords: AU-011; Belzupacap sarotalocan; Choroidal melanoma; Plaque radiotherapy; Matched case control; Visual acuity; bel-sar
MeSH Terms: conditions — Uveal Melanoma | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Patients with primary Choroidal Melanoma and Indeterminate Lesions who have received belzupacap sarotalocan (bel-sar; AU-011) in a previous Aura sponsored clinical trial
  Interventions: Drug: AU-011
- Control Group: Patients who are planned to receive plaque radiotherapy for the treatment of IL/CM based on the expert judgment of the investigator
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Patients who are planned to receive plaque radiotherapy for the treatment of IL/CM based on the expert judgment of the investigator
  Groups: Control Group
Drug: AU-011 — Previously received
  Other Names: belzupacap sarotalocan; bel-sar
  Groups: Case Group

SUMMARY:
This is a prospective multicenter, group-matched study of patients with primary indeterminate lesions or choroidal melanoma who receive treatment with belzupacap sarotalocan (bel-sar; AU-011) and patients who are planned to receive standard of care (SOC) treatment with plaque radiotherapy (plaque) to compare the visual outcomes of AU-011 and plaque radiotherapy.

DETAILED DESCRIPTION:
Up to approximately 45 patients who are planned to receive plaque radiotherapy for the treatment of IL/CM based on the expert judgment of the Investigator are planned to be enrolled.

ELIGIBILITY:
Have per the investigator's expert clinical judgment, a clinical diagnosis of primary indeterminate lesion or choroidal melanoma based on the clinical history, ophthalmic examination, fundus photography and conventional ocular ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary Choroidal Melanoma and Indeterminate Lesions who are planned to receive plaque radiotherapy (Control Group) and subjects with primary Choroidal Melanoma and Indeterminate Lesions who participated in previous Aura Biosciences sponsored clinical trial. (Case Group)
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 5 years
  Change from baseline in logMAR visual acuity score at 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Aura Biosciences, Inc.
Locations (7):
- United States (7):
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Oregon Health & Science University Casey Eye Institute, Portland, Oregon
  - Retina Consultants of Carolina, PA, Greenville, South Carolina
  - St. Thomas Health/Tennessee Retina, P.C., Nashville, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - University of Wisconsin Dept of Ophthalmology & Visual Sciences, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.aurabiosciences.com